CLINICAL TRIAL: NCT00674518
Title: Health Promotion Intervention: Sedentary Primary Care Patients
Brief Title: Changing Healthy Outcomes In Clinic Environments
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerry Kuehl, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1K23RR017554-01A2 (NIH)
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Physical Inactivity; Diabetes
Keywords: Health Promotion; Health Behavior Change; Physical Activity; Dietary Change; Weight Loss; Obesity
MeSH Terms: conditions — Obesity; Sedentary Behavior; Diabetes Mellitus; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling (Experimental): One-on-one sessions conducted by a professional motivational counselor to explore ways to help motivate participants to exercise, eat healthier, and lose weight.
  Interventions: Behavioral: One on one counseling
- Group (Experimental): A nutrition and exercise specialist will lead and teach a group of 4 to 5 subjects in healthy nutrition, exercise and weight loss habits
  Interventions: Behavioral: Group/team - based health education
- MD Advice (Active Comparator): A physician will provide exercise and nutrition advice to participants immediately following testing
  Interventions: Behavioral: PACE physician counseling

INTERVENTIONS:
Behavioral: One on one counseling — Motivational Interviewing
  Arms: Counseling
Behavioral: Group/team - based health education — peer led, scripted health promotion curriculum in groups of 4-5 individual, with team building activities and health education for 12, 1-hour sessions per year.
  Arms: Group
Behavioral: PACE physician counseling — PACE format for physician exercise and nutrition counseling annually.
  Arms: MD Advice

SUMMARY:
This study will compare three methods of counseling to determine which is most effective at motivating participants to adopt healthy lifestyle habits. The three methods are: individual counseling, working in groups with a health educator, and receiving advice from a physician. The health goals for subjects in this study are: 1) increase physical activity to 30 minutes each day, 2) reduce fat intake to less than 30% of total calories, 3) increase consumption of fruits and vegetables to at least 5 servings each day, and 4) reduce percentage of body fat to a healthy level.

DETAILED DESCRIPTION:
The benefits of physical activity and proper nutrition have been well established to prevent and reduce the devastating effects of chronic illness including, cardiovascular disease, diabetes, and obesity. Unfortunately, nearly 80% of individuals fail to get enough exercise and eat a proper diet to alter these health disorders. In the United States, physicians do not routinely counsel patients about physical activity and nutrition. Although few studies have examined promotion of physical activity in the primary care setting, most have been disappointing. Achieving and maintaining healthy behaviors remain a major challenge to promoting health and caring for illness. This research proposals aims are to a) evaluate two health behavior change intervention strategies to improve physical activity and dietary behaviors among sedentary patients in a primary care office; and b) assess by cost-benefit analysis, the impact of each model intervention. After initial recruitment from OHSU Internal Medicine and Family Practice clinics, 105 sedentary patients will be randomly assigned to Model 1, Model 2, or Model 3. Model #1, a one-on-one, individualized counseling intervention known as Motivational Interviewing, based on the transtheoretical model of behavior change, will use twelve health educator counseling meetings and ten bi-weekly follow-up phone calls the first year and six 60-minute sessions will occur in the second year of the intervention. Model #2, a team-centered intervention where the health promotion curriculum is delivered by a group facilitator to a team of patients (based on the social influence theory) consists of twelve 60-minute peer facilitated group meetings and ten follow-up phone calls, with six sessions occurring the second year of the full outcome study. Group facilitators will be trained and use scripted lesson plans. Model #3, a usual practice control condition (5 minute physician advice using the Physician Advice Counseling Exercise or PACE format). Models 1 and 2 contact hours are the same. Year 01 is the pilot study to revise and refine the curriculum and study protocol. The full intervention will last two years while the behavior change durability will be assessed over another full year. The study's primary outcomes are increased physical activity as measured by peak oxygen uptake and survey, dietary changes assessed by intake survey, and body composition changes as measured by DEXA. Secondary outcome measures include blood pressure lipid and lipoprotein levels, biochemical markers of inflammation (CRP) and hormonal markers of obesity. Outcomes will be assessed using repeated measures design. Relationships among mediators, the intervention, and the outcome measures will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patient patients who are sedentary (less than one exercise bout per week
* 30 - 65 years old
* In stable health, defined as an absence of serious chronic disease (i.e., recent myocardial infarction or CVA, uncontrolled metabolic conditions like thyrotoxicosis or poorly controlled diabetes mellitus).
* If the participants are taking medication for medical conditions, they have to be on a stable dose for at least three months with no medication change in past 3 months.
* Participants must be independent in living and able to obtain weekly transportation to OHSU
* able to increase their physical activity.

Exclusion Criteria:

* Non ambulatory
* Contraindications to exercise due to medical conditions using the AHA criteria and the ACSM Guidelines For Exercise Testing and Prescription. Examples are CAD, CHF, Recent CVA, poorly controlled DM (fasting glucose over 200 mg/dl), poorly controlled HTN, Severe COPD, Thyrotoxicosis, and Morbid Obesity with BMI > 40.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improve physical activity and dietary behaviors among sedentary patients | annually x 3 years

SECONDARY OUTCOMES:
Improve biomarkers of obesity including glucose, lipid levels, CRP, leptin and insulin. | annually x 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Kuehl KS, Elliot D, Edholm K, Frohnmayer S. Changing Healthy Outcomes In Clinical Environments (CHOICE) Study. Annals of Behavioral Medicine 33(Supplement):S094, 2007.